CLINICAL TRIAL: NCT06933277
Title: Observational Study on the Combination of Selinexor With Bortezomib and Dexamethasone (SVd) for the Treatment of Multiple Myeloma Patients
Brief Title: Observational Study on the Combination of Selinexor With Bortezomib and Dexamethasone for the Treatment of MM Patients
Status: Recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: MM0225
Record Dates: First submitted 2025-04-03; First posted 2025-04-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
Keywords: selinexor; bortezomib; dexamethasone
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study aiming at collecting efficacy and safety data on the use of SVd outside clinical trials, for the treatment of adult patients with MM who have received 1-3 prior line of therapy.

A minimum of 159 patients is required. Overall study duration is estimated in 36 months.

DETAILED DESCRIPTION:
This is a non-interventional, national, multicenter prospective and retrospective observational study aiming at collecting efficacy and safety data on the use of SVd outside clinical trials, for the treatment of adult patients with MM who have received 1-3 prior line of therapy.

All the sites participating in the study are using SVd in clinical practice. According to sample size calculation, a minimum of 159 patients is required.

Overall study duration is estimated in 36 months: 24 months on enrolment and at least 12 months of observation.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years old at the time of SVd initiation
* Signed informed consent (if applicable).
* Diagnosis of symptomatic MM, as defined by the International Myeloma Working Group (IMWG) criteria.
* Relapse after one to three lines of therapy.
* Treatment with SVd, (i.e., having already received at least one dose) at the time the combination has entered clinical practice in Italy (AIFA authorization)
* Prior treatment with and refractoriness to lenalidomide.

Exclusion Criteria:

- Previous exposure to selinexor.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: this study will include patients who will start SVD treatment during the study enrolment period or who received at least one dose of the treatment according to AIFA authorization before the study inclusion date.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
SdV therapy effectiveness in terms of Progression Free Survival | at 12 months
  to describe the effectiveness of the use of SVd therapy outside clinical trials in terms of Progression free survival after 12 months from the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elena Zamagni, Principal Investigator — UOC di Ematologia Policlinico S.Orsola AOU di Bologna
Locations (1):
- Aou Careggi - Sod Ematologia, Florence, Italy